CLINICAL TRIAL: NCT03646760
Title: The Improving ATTENDance to Cardiac Rehabilitation Trial
Acronym: iATTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steven J. Keteyian, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFHS iATTEND; R33HL143099 (NIH)
Record Dates: First submitted 2018-08-14; First posted 2018-08-24 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Heart Failure; Heart Valve Diseases; Cardiac Event; Angina Pectoris; Coronary Artery Disease
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Heart Valve Diseases; Cardiovascular Diseases; Angina Pectoris; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Cardiac Rehabilitation (HYCR) (Experimental)
  Interventions: Behavioral: HYCR
- Center Based cardiac Rehabilitation (CBCR) (Active Comparator)
  Interventions: Behavioral: CBCR

INTERVENTIONS:
Behavioral: HYCR — This group involves a hybrid design, with the frequency of center based cardiac rehabilitation (CBCR) visits and HYCR visits individualized and modified based on the subject's personal preferences and their family, transportation and work constraints. Patients in HYCR will engage in at least one CBCR visit. Patients will have the video app loaded to their smart phone or tablet (or that of a "willing to assist" family member or friend). HYCR patients receive a chest strap/wrist heart rate device to document HR before, during, and/or after exercise during the TM session. Program education for patients in HYCR will be delivered using the twenty-eight, 7-15 min audio PDF's that are free to access from the Health System's web site.
  Arms: Hybrid Cardiac Rehabilitation (HYCR)
Behavioral: CBCR — This group will attend 2-3 sessions of cardiac rehabilitation per week at the investigator's Detroit location. Program education for patients in CBCR will be delivered during eight. 1 hour education lectures taught by staff (exercise physiologists and registered dieticians).
  Arms: Center Based cardiac Rehabilitation (CBCR)

SUMMARY:
The benefits of cardiac rehabilitation are well known. However, despite center based cardiac rehabilitation (CBCR) representing guideline-based care for patients with cardiovascular disease, most patients do not complete the maximum number of sessions allowed by third party insurance payers. As such, many patients may not be receiving the full clinical benefit ascribed to CR. This study will assess the efficacy of an innovative approach to CR delivery on attendance by combining both center-based and remote- or home-based CR sessions. The intervention group combines center-based CR and remote-/home-based CR and is tailored to the individual needs of each patient, accomplished with the assistance of an easy-to-access telecommunications methodology (telemedicine)

ELIGIBILITY:
Inclusion Criteria:

1. Has agreed to participate in CR and has experienced a cardiac event (myocardial infraction, coronary revascularization, heart valve surgery, or cardiac transplant in the past 6 months; diagnosed with chronic, stable AHA/ACC stage B or C heart failure or Canadian class 0-2 stable angina pectoris)
2. Lives in or plans to remain in the greater Detroit, MI area for the next year
3. Age 18-85 years of age
4. Agrees to attend at least one CBCR session
5. Agrees to scheduling at least 2, up to 3, CR sessions (either CBCR or HYCR)/wk
6. Has demonstrated to research staff their ability to access and connect to the internet via smart phone or tablet and already has access to satisfactory home- or community-based exercise equipment

Exclusion Criteria:

1. Received a left ventricular assist device, receiving continuous inotropic support (e.g., milrinone), or undergoing hemodialysis
2. Angina at rest or with a low functional capacity (< 2 METs)
3. Advanced cancer, advanced risk for falling, limiting cognitive impairment, or other advanced disorder that limits participation in CR

   1. Advanced risk for falling will be assessed by 5X sit-to-stand test, with a cut-off score of >15 seconds
   2. Cognitive assessment will be completed using the Mini-Cog instrument, with a cut-off score < 3 used to exclude potential subjects.
4. Severe arrhythmia unless adequately treated (e.g., implantable cardiac defibrillator)
5. Pregnant or plan to become pregnant in the next year.
6. Major cardiovascular procedure or hospitalization planned in the next 6 months
7. Less than 12 month life expectancy
8. Participation in another clinical trial that interferes with iATTEND participation, follow-up, data collection, exercise capacity or quality of life.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Keteyian, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

REFERENCES:
- [Derived] Keteyian SJ, Grimshaw C, Ehrman JK, Kerrigan DJ, Abdul-Nour K, Lanfear DE, Brawner CA. The iATTEND Trial: A Trial Comparing Hybrid Versus Standard Cardiac Rehabilitation. Am J Cardiol. 2024 Jun 15;221:94-101. doi: 10.1016/j.amjcard.2024.04.034. Epub 2024 Apr 25. PMID 38670326
- [Derived] Keteyian SJ, Grimshaw C, Brawner CA, Kerrigan DJ, Reasons L, Berry R, Peterson EL, Ehrman JK. A Comparison of Exercise Intensity in Hybrid Versus Standard Phase Two Cardiac Rehabilitation. J Cardiopulm Rehabil Prev. 2021 Jan 1;41(1):19-22. doi: 10.1097/HCR.0000000000000569. PMID 33351540

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
Started | 142 | 140
Completed | 81 | 78
Not Completed | 61 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR) | Total
Number analyzed (Participants) | 142 | 140 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 68 | 154
  >=65 years | 56 | 72 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 97 | 94 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 76 | 76 | 152
  White | 62 | 59 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of CR Sessions Completed Within 6 Months in Patients Randomized to HYCR vs. Patients Randomized to Traditional CBCR (Usual Care).
Time Frame: Baseline to 6 months
Measure: Mean (Standard Error); unit: Number of cardiac rehab sessions
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
Number analyzed (Participants) | 142 | 140
Number of cardiac rehab sessions | 28.7 (11.8) | 27.6 (11.8)

2. Primary Outcome: Percentage of Patients Completing 36 CR Sessions Within 6 Months Among Patients Randomized to the HYCR Program vs. Patients Randomized to the CBCR Program.
Description: Outcome measure is the percent of people who complete all 36 CR sessions and the mean value reported represents the average percentage for all patients in both study groups.
Time Frame: Baseline to 6 months
Measure: Number; unit: % of patients completing 36 sessions
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
Number analyzed (Participants) | 142 | 140
% of patients completing 36 sessions | 58.5 | 50.7

3. Secondary Outcome: Improvement in Exercise Capacity, as Measured by Distance Walked During the Six Min Walk (6MW) Test, in Patients Randomized to HYCR vs Patients Randomized to CBCR.
Description: Improvement in exercise capacity was calculated as the change in distance from the start of cardiac rehab (T1) and within 1 week after the last CR session of a patient or 6 months after completing T1 (whichever came first).
Time Frame: Baseline to 6 months
Population: Analyses represent complete cases for Center Based Only CR and Hybrid CR
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
Number analyzed (Participants) | 108 | 105
Meters | 46 (46) | 50 (53)

4. Secondary Outcome: Improvement in Exercise Capacity, as Measured by Peak Oxygen Uptake (VO2), in Patients Randomized to HYCR vs Patients Randomized to CBCR.
Description: as for outcome 3
Time Frame: Baseline to 6 months
Population: Analyses represent complete cases for Center Based Only CR and Hybrid CR
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
Number analyzed (Participants) | 94 | 92
mL/kg/min | 2.3 (2.8) | 1.9 (2.8)

5. Secondary Outcome: Improvement in Quality of Life (QOL), as Measured by the Total Score for Dartmouth COOP, in Patients Randomized to HYCR vs Patients Randomized to CBCR.
Description: 5-point Likert-type scaling, with 1 being more positive and 5 being more negative. Lower scores indicate higher levels of quality of life.
  Improvement in qualify of life was calculated as the change in distance from the start of cardiac rehab (T1) and within 1 week after the last CR session of a patient or 6 months after completing T1 (whichever came first).
Time Frame: Baseline to 6 months
Population: Analyses represent complete cases for Center Based Only CR and Hybrid CR
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
Number analyzed (Participants) | 108 | 108
units on a scale | -3.9 (5.0) | -3.4 (5.3)

ADVERSE EVENTS:
Time Frame: 9-12 months, from the time patient enrolled into the study until they completed final study visit or 12 months from enrollment whichever came first.
Arm/Group | Hybrid Cardiac Rehabilitation (HYCR) | Center Based Cardiac Rehabilitation (CBCR)
All-Cause Mortality (participants affected / at risk) | 1/142 | 3/140
Serious Adverse Events (participants affected / at risk) | 1/142 | 0/140
Other Adverse Events (participants affected / at risk) | 8/142 | 3/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid Cardiac Rehabilitation (HYCR) (N=142) | Center Based Cardiac Rehabilitation (CBCR) (N=140)
Stroke (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid Cardiac Rehabilitation (HYCR) (N=142) | Center Based Cardiac Rehabilitation (CBCR) (N=140)
Unstable Angina (Cardiac disorders) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03646760/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03646760/ICF_001.pdf